CLINICAL TRIAL: NCT01428869
Title: The Effect of Combination Statin, Acetylsalicylic Acid and Dutasteride Use on Prostate Cancer - a Sub Analysis of the REDUCE Trial
Brief Title: Combination Statin, Acetylsalicylic Acid and Dutasteride Use in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1000AE
Record Dates: First submitted 2011-08-26; First posted 2011-09-05 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer
Keywords: Statins; acetylsalicylic acid; dutasteride; Prostate Cancer; Lower urinary tract symptoms; prevention; drug interactions
MeSH Terms: conditions — Prostatic Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Specimens were retained as part of the REDUCE protocol, but no biospecimens are required for the current protocol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- statin+ASA+dutasteride
- statin+ASA
- dutasteride+statin
- dutasteride+ASA

SUMMARY:
The purpose of this study is to assess whether there is any interaction between statins, acetylsalicylic acid (ASA) and dutasteride on protection from prostate cancer, the development of high grade prostate cancer, or lower urinary tract symptoms.

DETAILED DESCRIPTION:
A review of data collected from REDUCE (REduction by DUtasteride of prostate Cancer Events) study participants will be performed. Data required for the analysis includes: ethnicity, prostate specific antigen (PSA) levels, prostate volumes, presence of diabetes, concomitant medication use (for statin and ASA), prostate biopsy results at 2 and 4 years, body mass index (BMI), digital rectal exam (DRE) results, family history of Prostate Cancer and benign prostatic hyperplasia (BPH) outcomes: urinary retention, international prostate symptom score (IPSS), urinary tract infections (UTI)s.

The association of drug interactions with prostate cancer will be explored by using a multivariate logistic regression model including all possible interaction terms between dutasteride, ASA and statins (i.e. statin+ASA+dutasteride, statin+ASA, dutasteride+statin, dutasteride+ASA). Any interaction term found to be insignificant ( i.e. p>0.05) will be removed from the model. If a statistically significant interaction term is identified, the study cohort will be stratified by drug use, and the relative risk (RR)of prostate cancer among the different drug users will be reported. To control for potential confounders, a multivariate regression model will be constructed adjusting for age, family history of prostate cancer, DRE results and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received dutasteride or placebo and had at least one post-baseline prostate biopsy

Exclusion Criteria:

* Participants not taking concomitant statins or ASA

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants of the REDUCE trial (negative prostate biopsy at baseline) who had at least one post-baseline prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 8231 (Actual)
Dates: Start 2011-08; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Prostate Cancer | 4 years
  The relative risk of prostate cancer development in REDUCE study participants treated with a combination of statins, acetylsalicylic acid and dutasteride.

SECONDARY OUTCOMES:
Diagnosis of High Grade Prostate Cancer | 4 years
  The relative risk of high grade prostate cancer development in REDUCE study participants treated with a combination of statins, acetylsalicylic acid and dutasteride
Improvement of Lower Urinary Tract Symptoms | 4 years
  The impact of combination statin, acetylsalicylic acid and dutasteride use on lower urinary tract symptoms in REDUCE study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Fleshner, MD MPH FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada